CLINICAL TRIAL: NCT04712630
Title: Clinical and Radiographic Outcomes of the Apical Approach in Periodontal Surgery Reconstruction With and Without Graft Materials: Non-Incised Papillae Surgical Approach (NIPSA). A Randomized Controlled Clinical Trial
Brief Title: Non-Incised Papillae Surgical Approach (NIPSA) With and Without Graft
Acronym: NIPSAGRAFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Antonio José Ortiz Ruiz, MD, Professor and researcher, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2441/2019
Record Dates: First submitted 2021-01-14; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Periodontitis; Periodontal Diseases; Periodontal Pocket; Periodontal Attachment Loss
MeSH Terms: conditions — Periodontitis; Periodontal Diseases; Periodontal Pocket; Periodontal Attachment Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIPSA without grafting biomaterial (Experimental): A single horizontal or oblique apical incision will be made in the mucosa located on the bony cortex, far from the marginal tissues and apically to the edge of the bony crest delimiting the defect. The tissue coronal to the incision will be raised full thickness, trying to maintain the preoperative papillae architecture intact. The granulation tissue and epithelium of the pocket will be eliminated. The affected root will be scaled and planed, and calculus eliminated. Once the defect will be debrided, the enamel matrix derivates will be applied. Then the incision line will be sutured by a double suture line to facilitate closing without tension: The first with internal horizontal mattress sutures to approximate the connective tissue of both edges of the mucosal incision, and the second with single interrupted sutures.
  Interventions: Procedure: Non-incised papila surgical approach without grafting biomaterial
- NIPSA with grafting biomaterial (Active Comparator): A single horizontal or oblique apical incision will be made in the mucosa located on the bony cortex, far from the marginal tissues and apically to the edge of the bony crest delimiting the defect. The tissue coronal to the incision will be raised full thickness, trying to maintain the preoperative papillae architecture intact. The granulation tissue and epithelium of the pocket will be eliminated. The affected root will be scaled and planed, and calculus eliminated. Once the defect will be debrided, the enamel matrix derivates will be applied and the bone defect will be filled with a composite of xenograft and enamel matrix derivates. Then the incision line will be sutured by a double suture line to facilitate closing without tension: The first with internal horizontal mattress sutures to approximate the connective tissue of both edges of the mucosal incision, and the second with single interrupted sutures.
  Interventions: Procedure: Non-incised papila surgical approach with grafting biomaterial

INTERVENTIONS:
Procedure: Non-incised papila surgical approach without grafting biomaterial — Periodontal reconstructive surgery
  Arms: NIPSA without grafting biomaterial
Procedure: Non-incised papila surgical approach with grafting biomaterial — Periodontal reconstructive surgery
  Arms: NIPSA with grafting biomaterial

SUMMARY:
This study compared the clinical outcomes of the non-incised papila surgical approach (NIPSA) alone and with grafting biomaterial.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with periodontitis.
* plaque index and bleeding index of < 30%.
* periodontal lesions with pocket probing depth > 5 mm.
* intrabony defect > 3 mm.
* intrabony defect configuration including a 1 and/or 2-wall component, always involving the buccal wall.

Exclusion Criteria:

* patients with systemic diseases that contraindicated treatment.
* third molars.
* teeth with incorrect endodontic or restorative treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth (PD) | 12 months
  Probing pocket depth will be assessed with a periodontal probe, measured in mm from the gingival margin to the bottom of the pocket
Clinical attachment level (CAL) | 12 months
  Clinical attachment level will be assessed with a periodontal probe, measured in mm from the cementoenamel junction (CEJ) to the bottom of the pocket.
Recession (REC) | 12 months
  Recession, will be assessed with a periodontal probe, measured in mmm on the buccal aspect, from the CEJ to the gingival margin zenith.
Location of the tip of the papillae (TP) | 12 months
  Location of the tip of the papillae. Taking as reference the level of the mid-axis of the tooth, will be measured the distance from the CEJ at the zenith of the tooth to the tip of the papilla. A positive value will be recorded when the tip of the papillae is located coronally to the CEJ and a negative value otherwise.
  This outcome will be assessed with a periodontal probe and measured in mm.
Keratinized tissue width (KT) | 12 months
  Keratinized tissue width will be assessed with a periodontal probe, measured in mm on the buccal aspect, from the gingival margin to the mucogingival line.
Bleeding on probing | 12 months
  Bleeding on probing could be positive or negative.

SECONDARY OUTCOMES:
Supra-alveolar attachment gain (SUPRA-AG) | 12 months
  Subtracting the 12-month CAL from the intra-surgically BC-CEJ will provide the SUPRA-AG result.
Wound closure (WC) | 1 week
  Complete wound closure (CWC = 2) Incomplete wound closure (IWC = 1) necrosis (NT = 0).

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Odontologico Del Sureste Slp, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreno Rodriguez JA, Caffesse RG. Nonincised Papillae Surgical Approach (NIPSA) in Periodontal Regeneration: Preliminary Results of a Case Series. Int J Periodontics Restorative Dent. 2018;38(Suppl):s105-s111. doi: 10.11607/prd.3195. PMID 30118534
- [Background] Moreno Rodriguez JA, Ortiz Ruiz AJ, Caffesse RG. Periodontal reconstructive surgery of deep intraosseous defects using an apical approach. Non-incised papillae surgical approach (NIPSA): A retrospective cohort study. J Periodontol. 2019 May;90(5):454-464. doi: 10.1002/JPER.18-0405. Epub 2018 Nov 28. PMID 30421495
- [Background] Moreno Rodriguez JA, Ortiz Ruiz AJ, Caffesse RG. Supra-alveolar attachment gain in the treatment of combined intra-suprabony periodontal defects by non-incised papillae surgical approach. J Clin Periodontol. 2019 Sep;46(9):927-936. doi: 10.1111/jcpe.13158. Epub 2019 Jul 22. PMID 31190409
- [Derived] Moreno Rodriguez JA, Ortiz Ruiz AJ. Apical approach in periodontal reconstructive surgery with enamel matrix derivate and enamel matrix derivate plus bone substitutes: a randomized, controlled clinical trial. Clin Oral Investig. 2022 Mar;26(3):2793-2805. doi: 10.1007/s00784-021-04256-1. Epub 2021 Nov 17. PMID 34791548